CLINICAL TRIAL: NCT05305833
Title: Stem Cells Transplantation for Temporomandibular Joint Disease: Phase I/II Study
Brief Title: Stem Cells and Stromal Vascular Fraction for Temporomandibular Joint Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Zeynep Burcin GONEN, Associate Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021/584
Record Dates: First submitted 2021-11-12; First posted 2022-03-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Temporomandibular Joint Disorders; Temporomandibular Disorder; Temporomandibular Joint Osteoarthritis; Temporomandibular Joint Pain; Temporomandibular Joint Effusion
MeSH Terms: conditions — Temporomandibular Joint Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- umbilical cord derived mesenchymal stem cells transplantation group (Experimental): taking umbilical cord derived mesenchymal stem cells
  Interventions: Biological: Stem Cells
- stromal vascular fraction cells application group (Experimental): taking stromal vascular fraction cells
  Interventions: Biological: Stem Cells

INTERVENTIONS:
Biological: Stem Cells — ATMP

SUMMARY:
It will be evaluate the safety of mesenchymal stem cells and adipose tissue derived stromal vascular fraction (SVF) in temporomandibular joint disease cases.

DETAILED DESCRIPTION:
umbilical cord derived mesenchymal stem cells produced under GMP facility in Erciyes University and SVF produced in operation theatre.

ELIGIBILITY:
Inclusion Criteria:

* Chronic temporomandibular arthritic disorder
* History of pain and joint noises for at least 3 months
* Must have more than VAS 5 TMJ pain
* must have internal derangement of TMJ
* Limited mouth opening
* Magnetic resonance imaging evidence of effusion or degeneration
* Already treated with conservative methods (occlusal splint,pharmacological and/or physio-kinesio therapy) without satisfactory benefit.

Exclusion Criteria:

* Cancer patients
* Immunosupressed patients
* Previous TMJ traumas and fractures
* Previous TMJ surgeries
* TMJ ankylosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Pain at 15th day | 15th day
  using by Visual Analogue Scale (VAS); higher scores mean worse outcome
Change from baseline maximum mouth opening at 15th day | 15th day
  the distance between incisal edge of maxillary central incisor to the incisal edge of mandibular central incisor, when the mouth is opened as wide as possible painlessly
Change from baseline maximum mouth opening at 1 month | 1. month
  the distance between incisal edge of maxillary central incisor to the incisal edge of mandibular central incisor, when the mouth is opened as wide as possible painlessly at first month; higher scores means a better outcome
Change from baseline maximum mouth opening at 3 months | 3. month
  the distance between incisal edge of maxillary central incisor to the incisal edge of mandibular central incisor, when the mouth is opened as wide as possible painlessly at third month; higher scores means a better outcome
Change from baseline maximum mouth opening at 6 months | 6. month
  the distance between incisal edge of maxillary central incisor to the incisal edge of mandibular central incisor, when the mouth is opened as wide as possible painlessly at 6th month,higher scores means a better outcome
Change from baseline pain at 1 month | 1. month
  using by Visual Analogue Scale (VAS)
Change from baseline pain at 3 month | 3. month
  using by Visual Analogue Scale (VAS)
Change from baseline pain at 6 month | 6. month
  using by Visual Analogue Scale (VAS) higher scores mean worse outcome

SECONDARY OUTCOMES:
Change from baseline 'comfort ' at 6th month | 6 months
  using by Visual Analogue Scale (VAS); higher scores mean better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep B Gonen, DDS,PHD, Principal Investigator — Assoc.Prof
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)